CLINICAL TRIAL: NCT03940937
Title: Cadence and Intensity in Adults With Type 2 Diabetes
Acronym: CADENCE-T2DM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Stuart R Chipkin, Research Professor, University of Massachusetts, Amherst
Other Study IDs: CADENCE-T2DM
Record Dates: First submitted 2018-09-11; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Type 2 Diabetes Mellitus; Walking
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to measure and link cadence (number of steps taken in a minute) to intensity of physical activity (e.g., low-intensity, moderate intensity, vigorous-intensity) in adults (40- 65 years-old) with type 2 diabetes.

DETAILED DESCRIPTION:
There will be up to two lab visits for participants, all of which will be completed in the Physical Activity and Health Lab at University of Massachusetts Amherst (consent, physical examination and entire research protocol, 2.5-3.5 hrs for all participants).

The first visit will consist of an orientation session. This orientation will begin with screening questions to determine eligibility and obtaining informed consent (45 min), followed by a physical exam and resting ECG for all participants (30 min):

Screening Questions: Participants will self-report their diagnosis of type 2 diabetes and year of diagnosis. Medication used for controlling diabetes will be determined by participants bringing their medication bottle or a photo of its label. Participants will answer additional questions (documentation attached) in an interview-style format with research staff to determine eligibility (15 min). These questions will be derived from the American Heart Association's (AHA) risk stratification found in the 2013 edition of the American College of Sports Medicine's (ACSM's) Resource for The Health Fitness Specialist. According to this screening, all participants with type 2 diabetes are considered high risk but the additional cardiac, pulmonary, and metabolic disease-related questions will be used for descriptive purposes. Given the low impact of this protocol, the volunteer's personal physician does not need to provide clearance. The PI, who is a physician, will be available to review individual circumstances prior to testing.

Informed Consent: Research staff will present an orientation slideshow to participants regarding the study purpose, study procedures, and rights as a participant (slideshow attached). Participants will then review and sign informed consent documents. (30 min)

Physical Exam: A physical exam will be conducted by study staff under the guidance of the medical director (Stuart Chipkin, MD) to assess for medical conditions that may interfere with the exercise protocol and ensure participant safety. In addition, the medical director will conduct tests for diabetic neuropathy with the neuropathy symptom and change (NSC) score, neuropathy impairment score (NIS). The NSC consists of a series of questions about neuropathy-related pain and numbness, maneuvers that relieve symptoms, and arousal from sleep. The NIS is a battery of tests that assess the ankle reflex as well as vibration, pin-prick, and temperature sensation in the great toes. (15 min)

Electrocardiogram (ECG). A resting 12-lead electrocardiogram will be performed and reviewed by the medical director prior to the exercise protocol (15 min).

Metabolic testing will then occur during the same session or a second study visit. All testing will be overseen by trained study staff with an MS or PhD in Exercise Science/Physiology or BS in Kinesiology as well as the medical director. These accommodations meet the ACSM and AHA criteria for exercise protocols. Because responses to exercise are affected by 4 hr pre-exercise food intake participants will have fasted for 4 hrs prior to testing. The metabolic testing session will be comprised of anthropometric and demographic information collection, instrument attachment, blood glucose measurement, and treadmill walking:

Anthropometrics and demographic information collection: Measures will be taken of height, seating height, body mass, body fat percentage, BMI, and waist circumference. Questions will be asked to ascertain date of birth, gender, and race/ethnicity.

Instrument attachment: Non-invasive pedometers and accelerometers will be worn by participants to measure/monitor movement during treadmill testing. The purpose of attaching these devices is to test the criterion-validity of step-counting wearable devices during treadmill walking in adults with T2DM, and compare the results to those observed with healthy adults. This is a secondary aim of the study. Participants will also be fitted with a mobile indirect calorimeter (facemask and back harness) and chest strap heart-rate monitor for measuring oxygen consumption and heart-rate.

Blood glucose measurements: The medical investigator will check fingerstick glucose values using a standard FDA-approved glucose meter before and 30 minutes after completion of treadmill testing. Following guidelines from the American Diabetes Association (Colberg SR et al; Diabetes Care 2016; 39:2065-2079. DOI: 10.2337/dc16-1728), any subject with a pre-test blood glucose < 70 mg/dl will be given 15-20 grams of carbohydrate. For glucose values between 70-150 mg/dl, study staff will administer 0.5 grams of carbohydrate per kg body mass. In addition, the medical investigator will test glucose values at any point during the protocol that a participant reports symptoms of hypoglycemia (low blood sugar) such as feeling sweaty, shaky, or weak. Subjects will be given a light snack after the testing session and informed about the potential for low blood sugars following exercise. The light snack will consist of 15-20g of simple carbohydrates or glucose.

Treadmill walking: Throughout the treadmill walking protocol, ambulatory monitoring of ECG and blood pressure will be conducted for ensuring participant safety Participants will complete a series of 5-min bouts of treadmill walking. The first bout will be performed at 0.5 mph, with concurrent bouts increasing in 0.5 mph increments, and the test will be terminated upon participant or researcher volition or completion of the first bout when the participant 1) naturally selects to run instead of walk, 2) achieved 75% of their predicted maximum heart rate, or 3) reported a Borg Rate of Perceived Exertion Scale (see attachment document ) > 13, or 4) reaches a speed of 6.0 mph. Each bout will be separated by 2-5min of standing rest on the stopped treadmill. Participants will not be seated during the resting period, as this is a submaximal protocol and fatigue preventing its continuation and requiring seated rest would be an indication to end the test.

During treadmill testing, cadence (steps/min) will be assessed by the number of directly-observed steps divided by bout duration. Redundant video recording of the participant's feet will be conducted during the entirety of treadmill testing as a back-up method to confirm step counts. Indirect calorimetry will concurrently be used to measure oxygen uptake.

ELIGIBILITY:
Inclusion Criteria:

* Able to ambulate on a treadmill (self-reported)
* Diagnosed with type 2 diabetes (self-reported)
* Self-report participating in less than 30 minutes of moderate intensity exercise per day for most days of the week
* Able to fast for at least 4 hours prior to study visit involving the treadmill protocol
* Self-report having an HbA1c measure greater than 7% in the past 6 months

Exclusion Criteria:

* BMI - <18.5kg/m² or >40kg/m²
* Tobacco use - Currently a smoker or have smoked tobacco within the past 6 months.
* Insulin - Those with type 2 diabetes being controlled with insulin
* Ambulatory ability - Since the focus herein is on ambulatory activities, participants who use wheelchairs or other impairments that prevent normal ambulation will be excluded. This criterion is similar to that used by NHANES when selecting individuals (up to 85 years of age) to wear motion sensors.
* Resting Blood Pressure - Systolic blood pressure greater than 159 mmHg or diastolic blood pressure greater than 99mmHg
* Abnormal resting ECG (evaluated by physician) will be advised to see personal physician (participant provided with resting ECG results)
* Any condition/medication that may affect heart rate response to exercise testing.
* Current participation in any other study protocol which involves taking an experimental medication
* Hospitalization for mental illness within the past 5 years.
* Previous history of, or clinical symptoms or signs of, cardiovascular disease, stroke or transient ischemic attacks (TIAs), chest pain, unusual dyspnea during physical activity/ exercise, severe ankle edema, or intermittent claudication.
* Previous history of musculoskeletal injuries or problems causing severe pain during physical activity or exercise which interferes with daily activities.
* Participant experiences dizziness or balance impairment at rest or with exercise
* Participant is currently treated for kidney disease with dialysis, or has severe liver damage? (e.g., liver cirrhosis)
* Participant has a pacemaker or other implanted medical device (including metal joint replacements).
* Participant has chronic lung problems that make it difficult to breathe (e.g., Chronic Respiratory Diseases, Cystic Fibrosis, chronic obstructive pulmonary disease [COPD] or uses supplemental O2)
* Participant has Cancer treated with chemotherapy that affects breathing or heart rate
* Participant experiences shortness or breath at rest or during mild exertion
* Participant is pregnant.
* Participant is unable to complete all testing within a maximal two-week period
* Individuals wearing a full beard may need to be excluded from the study, as large amounts of facial hair around the mouth and nose interfere with the seal of the device that measures the air being breathed. Because of this we are seeking participants that are clean shaven or with a beard where areas around the nose and mouth are clean shaven (e.g. goatee).
* Any significant medical condition that may interfere with the study.

Ages: 40 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A convenience sample from the surrounding community consisting of twenty 40-65 yr old adults (10 men, 10 women) with pharmacologically-controlled type 2 diabetes (not using insulin). Participants must self-report being non-active (less than 30 minutes of moderate intensity exercise per day for most days of the week) and to have an HbA1c not at goal (therefore >7%) in the past 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Cadence (steps/min) | Through completion of the treadmill walking protocol that occurs during the study visit (approximately 1 hour)
  Cadence (steps/min) as assessed by direct observation of steps (hand-tallied counts) divided by time
Oxygen consumption (VO2; mL/kg/min) | Through completion of the treadmill walking protocol that occurs during the study visit (approximately 1 hour)
  The amount of oxygen consumed, as measured with indirect calorimetry, expressed per unit of body mass

CONTACTS AND LOCATIONS:
Overall Officials: Stuart C Chipkin, MD, Principal Investigator — University of Massachusetts Amherst, Department of Kinesiology
Locations (1):
- Totman Building, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tudor-Locke C, Rowe DA. Using cadence to study free-living ambulatory behaviour. Sports Med. 2012 May 1;42(5):381-98. doi: 10.2165/11599170-000000000-00000. PMID 22462794
- [Background] Caron N, Peyrot N, Caderby T, Verkindt C, Dalleau G. Energy Expenditure in People with Diabetes Mellitus: A Review. Front Nutr. 2016 Dec 22;3:56. doi: 10.3389/fnut.2016.00056. eCollection 2016. PMID 28066773
- See also: UMass Physical Activity and Health Lab — http://blogs.umass.edu/pahl/